CLINICAL TRIAL: NCT01801059
Title: Patient Activation To Increase Colon Cancer Screening (THE CHAT STUDY)
Brief Title: Patient Activation Intervention in Improving Screening Rates for Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Mira Katz, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: OSU-07104; NCI-2012-01922 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: colon cancer; Colorectal Cancer Screening
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I education CRC and CRC screening (Active Comparator): Educational intervention: Patients receive CRC and CRC screening information from an educational video and received a brochure focused on healthy hints to prevent CRC. Questionnaire administration prior to and after the intervention.
  Interventions: Other: educational intervention; Other: questionnaire administration
- Arm II education and patient activation intervention (Experimental): Educational intervention administered: Patients receive patient activation intervention comprising CRC and CRC screening information and communication skills training intervention by educational video and brochure, and they also receive a brochure focused on healthy hints to prevent CRC. Questionnaire administration prior to and after the intervention.
  Interventions: Other: educational intervention; Other: questionnaire administration

INTERVENTIONS:
Other: educational intervention — Receive patient activation intervention by educational video and brochure
  Other Names: intervention, educational
Other: educational intervention — Receive patient activation intervention by educational video
  Other Names: intervention, educational
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized clinical trial focused on activating the patient to ask their health care provider for a colorectal cancer screening test to improve screening rates for colorectal cancer. The patient activation intervention may increase information seeking, number of screening tests ordered and number of completed screening tests for colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test a patient activation intervention to improve colorectal cancer (CRC) screening rates using fecal occult blood test (FOBT) among male and female patients 50 years and older from the East Central Columbus Neighborhood Health Center.

SECONDARY OBJECTIVES:

I. To assess if there is a change in knowledge and attitudes about CRC screening after watching the educational video.

II. To assess the effectiveness of providing communication skills training for improving discussion focusing on CRC screening during the patient-provider visit.

OUTLINE: Patients are randomized to 1 of 2 arms prior to a medical visit.

ARM I (Education only): Patients receive CRC and CRC screening information by an educational video and a brochure with healthy hints to prevent CRC.

ARM II (Education and patient activation): Patients receive CRC and CRC screening information and communication skills training (patient activation) intervention by educational video and brochure and a brochure about healthy hints to prevent CRC.

After the medical visit, patients' medical records are reviewed at 1 month and 2 months after the visit to document CRC screening completion.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 50+ years of age
* Patient is in need of CRC screening
* Patient is in good health (e.g. no contraindications to having CRC screening, such as a history of colorectal cancer, congenital heart failure, renal failure, dialysis, dementia, severe arthritis, etc.)
* Patient is not pregnant
* Patient is able to speak, read, and understand English

Exclusion Criteria:

* Patient is within CRC screening guidelines
* Patient is at high risk for CRC
* Patient cannot understand English
* Patient cannot complete a CRC screening test

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2007-09; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Completion rate of CRC screening | Up to 2 months
  A test of two proportions will be used. If the two groups are different at baseline with respect to key covariates, then a logistic regression model will be used to assess the effect of the intervention on CRC screening controlling for possible confounding variables. The variables that differ between the two groups will be tested as confounders using risk-factor modeling. Summary statistics will be used to describe the time point that subjects receive CRC screening, either after the medical visit or after telephone barriers counseling, and relevant comparisons made.

CONTACTS AND LOCATIONS:
Overall Officials: Mira Katz, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu